CLINICAL TRIAL: NCT02820233
Title: Isolation and Characterization of ERBB Expressing Human Heart Progenitor Cells
Brief Title: Studies of Neuregulin/ERBB Signaling in Human Heart
Status: Recruiting | Type: Observational
Sponsor: Douglas B. Sawyer (Other)
Collaborators: MaineHealth (Other)
Responsible Party: Sponsor-Investigator, Douglas B. Sawyer, Chief Academic Officer, MaineHealth
Organization: MaineHealth (Other)
Other Study IDs: 4590
Record Dates: First submitted 2016-06-27; First posted 2016-06-30 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2024-07

CONDITIONS: Heart Disease; Vascular Disease; Heart Failure
MeSH Terms: conditions — Heart Diseases; Vascular Diseases; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, circulating monocytes, and cardiac tissue.
Oversight: Data Monitoring Committee: Yes | US Export: No

SUMMARY:
This study examines the role of the epidermal growth factor (EGF) receptor family and the EGF family of ligands in the regulation of non-myocytes isolated from the human heart.

DETAILED DESCRIPTION:
The EGF family of receptor tyrosine kinases (a.k.a. ERBB receptors) mediate the effects of the epidermal growth factor (EGF) family including Neuregulin-1β (NRG). NRG and ERBB1-4 are critical for cardiac development and maintenance of the adult heart. Current understanding of the role of EGF/NRG/ERBB signaling in the cardiovascular system is rapidly evolving due to recent findings in non-myocyte cell populations. This study is examining a population of progenitor cells in the adult human heart that responds to EGF and NRG. Subjects are enrolled who are scheduled to undergo heart surgery and are willing to allow for a small biopsy to be taken from their hearts during surgery. Biopsies are taken to the laboratory where cells are separated and analyzed by flow cytometry and grown in cell culture to understand how their biology is regulated by NRG and EGF.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of severe coronary artery disease scheduled to undergo coronary artery bypass surgery.

Exclusion Criteria:

* less than 18 years of age
* unwilling or unable to provide informed consent
* known active myocarditis
* hypertrophic cardiomyopathy
* constrictive pericarditis or other significant pericardial disease
* severe pulmonary hypertension
* significant renal impairment (Cr > 2.5 mg/dL)
* severe ventricular arrhythmias
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with coronary artery disease with scheduled coronary artery bypass surgery.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
The number of highly proliferative clones isolated | up to 14 days from isolation

SECONDARY OUTCOMES:
Flow cytometric ERBB receptor expression in highly proliferative clones isolated from heart tissue | up to 14 days from isolation

CONTACTS AND LOCATIONS:
Locations (1):
- Maine Medical Center, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Ryzhov S, Robich MP, Roberts DJ, Favreau-Lessard AJ, Peterson SM, Jachimowicz E, Rath R, Vary CPH, Quinn R, Kramer RS, Sawyer DB. ErbB2 promotes endothelial phenotype of human left ventricular epicardial highly proliferative cells (eHiPC). J Mol Cell Cardiol. 2018 Feb;115:39-50. doi: 10.1016/j.yjmcc.2017.12.013. Epub 2017 Dec 29. PMID 29291395
- [Background] Robich M, Ryzhov S, Kacer D, Palmeri M, Peterson SM, Quinn RD, Carter D, Sheppard F, Hayes T, Sawyer DB, Rappold J, Prudovsky I, Kramer RS. Prolonged Cardiopulmonary Bypass is Associated With Endothelial Glycocalyx Degradation. J Surg Res. 2020 Jul;251:287-295. doi: 10.1016/j.jss.2020.02.011. Epub 2020 Apr 30. PMID 32199337
- [Background] de Kay JT, Carver J, Shevenell B, Kosta AM, Tsibulnikov S, Certo E, Sawyer DB, Ryzhov S, Robich MP. Decreased expression of ErbB2 on left ventricular epicardial cells in patients with diabetes mellitus. Cell Signal. 2022 Aug;96:110360. doi: 10.1016/j.cellsig.2022.110360. Epub 2022 May 21. PMID 35609807